CLINICAL TRIAL: NCT00546078
Title: Safety and Immunogenicity Study of an Additional Dose of HPV Vaccine (580299) in Young, Adult Women in North America.
Brief Title: Follow-up Study to Evaluate the Safety and Immunogenicity of a HPV Vaccine (580299) in North America
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109628
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Results first posted 2009-12-15 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-10

CONDITIONS: Infections, Papillomavirus
Keywords: HPV vaccine; Cervical cancer; Human papillomavirus infection
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (2):
- Cervarix™ 4-Dose Group (Experimental): Subjects who had received 3 doses of Cervarix™ in study 580299/001 (NCT00689741), received a 4th dose of Cervarix™ on Day 0 in the current study.
  Interventions: Biological: Cervarix™
- Cervarix™ 3-Dose Group (Experimental): Subjects who had received 3 doses of placebo in study 580299/001 (NCT00689741), received 3 doses of Cervarix™ (Day 0, Month 1 and Month 6) in the current study.
  Interventions: Biological: Cervarix™

INTERVENTIONS:
Biological: Cervarix™ — Intramuscular injection, one or three doses
  Other Names: GSK Biologicals' HPV Vaccine GSK580299

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. This study will further evaluate induction of immune memory and anamnestic responses in women who previously took part in the primary study (580299/001) and follow-up study (580299/007). Subjects were aged 15-25 yrs at the time of entry into the primary study and participation in the follow-up study lasted approximately 6 years. In the primary and follow-up studies, subjects were protected against HPV-16 and HPV-18 endpoints and had sustained antibody responses to both vaccine types over at least 5.5 years of follow-up. All subjects from North American study sites that completed the follow-up study will be invited to take part in the current study. The study will evaluate the safety and immunogenicity of a dose of GSK Biologicals HPV vaccine (580299) in women who had been immunologically primed in the primary study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A subject whom the investigator believes that she can and will comply with the requirements of the protocol
* Must have received three doses of study vaccine or placebo control in study 580299/001.
* Must have completed study 580299/007.
* Written informed consent must be obtained from the subject prior to enrollment in the study.
* Healthy subjects, as established by medical history and history-directed clinical examination before entering into the study.
* Subject must have a negative urine pregnancy test.
* Subject must be at least three months post-termination of a pregnancy.
* Subject must be of non-childbearing potential,or subjects are required to be abstinent or use adequate contraceptive precautions for 30 days prior to vaccination. Subjects are also required to agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or breastfeeding.
* A woman planning to become pregnant or planning to discontinue contraceptive precautions during the study until approximately 2 months after the last vaccination.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned administration during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of each dose of vaccine. Administration of some routine vaccines up to 8 days before each dose of study vaccine is allowed.
* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* previous administration of components of the investigational vaccine outside of protocol 580299/001.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines,
* Hypersensitivity to latex
* Acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Cancer or autoimmune disease under treatment.
* Administration of immunoglobulins and/or any blood products within the three months (90 days) preceding enrollment or planned administration during the study period.
* Acute disease at the time of enrollment. All vaccines can be administered to persons with a minor illness
* Heavy bleeding or heavy vaginal discharge in which a pelvic exam cannot be performed.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2008-01-14; Primary Completion 2008-12-22 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (13):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Grove City, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- Canada (4):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Moscicki AB, Wheeler CM, Romanowski B, Hedrick J, Gall S, Ferris D, Poncelet S, Zahaf T, Moris P, Geeraerts B, Descamps D, Schuind A. Immune responses elicited by a fourth dose of the HPV-16/18 AS04-adjuvanted vaccine in previously vaccinated adult women. Vaccine. 2012 Dec 17;31(1):234-41. doi: 10.1016/j.vaccine.2012.09.037. Epub 2012 Oct 11. PMID 23063422
- [Background] Moscicki B et al. Anamnestic response elicited by a fourth dose of the HPV-16/18 ASO4-adjuvanted vaccine in young women. Abstract presented at European Research Organization on Genital Infection and Neoplasia 2010 (EUROGIN). Monte Carlo, Monaco, 17-20 February 2010.
- [Background] Moscicki B et al. Anamnestic response to non-vaccine types elicited by a fourth dose of the HPV-16/18 ASO4-adjuvanted vaccine in young women. Abstract presented at European Research Organization on Genital Infection and Neoplasia 2010 (EUROGIN). Monte Carlo, Monaco, 17-20 February 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject that enrolled into the study was not vaccinated and as such not reported as started in the participant flow.
Period: Overall Study
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Started | 65 | 50
Month 18 | 61 | 45
Completed | 61 | 43
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group | Total
Number analyzed (Participants) | 65 | 50 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (2.82) | 27.0 (2.89) | 27.5 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 50 | 115
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-human Papilloma Virus-16 (Anti-HPV-16) and Anti-HPV-18 Antibody Titers Greater Than or Equal to Pre-defined Cut-off Values
Description: Cut-off values assessed include 8 Enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: At Day 7 and Month 1 (Day 30)
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 61 | 45
Participants
  Anti-HPV-16 at Day 7 | 61 | 30
  Anti-HPV-16 at Month 1: number analyzed (Participants) | 57 | 45
  Anti-HPV-16 at Month 1 | 57 | 45
  Anti-HPV-18 at Day 7 | 61 | 26
  Anti-HPV-18 at Month 1: number analyzed (Participants) | 57 | 45
  Anti-HPV-18 at Month 1 | 57 | 45

2. Primary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) calculated on all subjects.
Time Frame: At Day 7 and at Month 1 (Day 30)
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 61 | 45
titer
  anti-HPV-16 Day 7 | 5894.9 [4734.0 to 7340.7] | 67.9 [27.2 to 169.7]
  anti-HPV-16 Month 1: number analyzed (Participants) | 57 | 45
  anti-HPV-16 Month 1 | 15410.7 [12807.9 to 18542.4] | 1231.1 [709.6 to 2135.9]
  anti-HPV-18 Day 7 | 3916.2 [3087.7 to 4967.0] | 20.7 [10.2 to 42.2]
  anti-HPV-18 Month 1: number analyzed (Participants) | 57 | 45
  anti-HPV-18 Month 1 | 8362.7 [6930.4 to 10091.1] | 442.0 [269.8 to 724.3]

3. Secondary Outcome: Number of Subjects With Anti-HPV-16 and Anti-HPV-18 Greater Than or Equal to Pre-defined Cut-off Values
Description: Cut-off values assessed include 8 EL.U/mL for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: At Month 7 and Month 18
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 55 | 43
Participants
  Anti-HPV-16 at Month 7 | 55 | 43
  Anti-HPV-16 at Month 18: number analyzed (Participants) | 49 | 40
  Anti-HPV-16 at Month 18 | 49 | 40
  Anti-HPV-18 at Month 7 | 55 | 43
  Anti-HPV-18 at Month 18: number analyzed (Participants) | 49 | 40
  Anti-HPV-18 at Month 18 | 49 | 40

4. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Titers
Description: Titers are given as GMTs calculated on all subjects.
Time Frame: At Month 7 and Month 18
Population: Analysis was performed on the APT cohort for immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 55 | 43
titer
  Anti-HPV-16 at Month 7 | 5826.9 [4742.4 to 7159.5] | 7166.5 [5954.3 to 8625.5]
  Ant-HPV-16 at Month 18: number analyzed (Participants) | 49 | 40
  Ant-HPV-16 at Month 18 | 3936.6 [3128.7 to 4953.1] | 1626.9 [1252.4 to 2113.5]
  Anti-HPV-18 at Month 7 | 2940.3 [2385.0 to 3625.0] | 3584.3 [2913.9 to 4408.9]
  Ant-HPV-18 at Month 18: number analyzed (Participants) | 49 | 40
  Ant-HPV-18 at Month 18 | 1802.5 [1407.9 to 2307.6] | 520.1 [382.9 to 706.4]

5. Secondary Outcome: Number of Subjects With Antibody Titers Against Other Oncogenic HPV Types (HPV-31 & HPV-45) Greater Than or Equal to 59 EL.U/mL
Time Frame: Day 0, Month 1 (Day 30), Month 7 and Month 18
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 61 | 45
Participants
  anti-HPV-31 Day 7 | 61 | 20
  anti-HPV-31 Month 1: number analyzed (Participants) | 58 | 45
  anti-HPV-31 Month 1 | 58 | 31
  anti-HPV-31 Month 7: number analyzed (Participants) | 55 | 43
  anti-HPV-31 Month 7 | 55 | 43
  anti-HPV-31 Month 18: number analyzed (Participants) | 49 | 40
  anti-HPV-31 Month 18 | 48 | 35
  anti-HPV-45 Day 7 | 61 | 18
  anti-HPV-45 Month 1: number analyzed (Participants) | 58 | 45
  anti-HPV-45 Month 1 | 58 | 32
  anti-HPV-45 Month 7: number analyzed (Participants) | 55 | 43
  anti-HPV-45 Month 7 | 55 | 43
  anti-HPV-45 Month 18: number analyzed (Participants) | 49 | 40
  anti-HPV-45 Month 18 | 49 | 35

6. Secondary Outcome: Anti-HPV-31 and Anti-HPV-45 Antibody Titers
Description: Titers are given as geometric mean titers (GMTs) calculated on all subjects.
Time Frame: Day 7, Month 1 (Day 30), Month 7 and Month 18
Population: Analysis was performed on the ATP cohort for immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 61 | 45
titer
  anti-HPV-31 Day 7 | 2075.3 [1635.4 to 2633.6] | 90.7 [55.8 to 147.4]
  anti-HPV-31 Month 1: number analyzed (Participants) | 58 | 45
  anti-HPV-31 Month 1 | 3705.8 [2902.4 to 4731.5] | 192.1 [110.7 to 333.4]
  anti-HPV-31 Month 7: number analyzed (Participants) | 55 | 43
  anti-HPV-31 Month 7 | 1193.8 [879.6 to 1620.2] | 878.3 [641.2 to 1202.9]
  anti-HPV-31 Month 18: number analyzed (Participants) | 49 | 40
  anti-HPV-31 Month 18 | 667.0 [470.2 to 946.3] | 225.4 [147.9 to 343.6]
  anti-HPV-45 Day 7 | 2347.7 [1869.9 to 2905.6] | 76.4 [49.9 to 116.9]
  anti-HPV-45 Month 1: number analyzed (Participants) | 58 | 45
  anti-HPV-45 Month 1 | 4491.5 [3655.6 to 5518.5] | 189.9 [113.6 to 317.4]
  anti-HPV-45 Month 7: number analyzed (Participants) | 55 | 43
  anti-HPV-45 Month 7 | 1503.1 [1149.7 to 1965.0] | 981.0 [778.6 to 1236.0]
  anti-HPV-45 Month 18: number analyzed (Participants) | 49 | 40
  anti-HPV-45 Month 18 | 890.2 [663.6 to 1194.1] | 185.1 [129.5 to 264.5]

7. Secondary Outcome: Number of Subjects With Cluster of Differentiation 4 (CD4) T Cell-mediated Immune Responses Specific to Defined Oncogenic HPV Types
Description: CD4 T cell-mediated immune responses against the antigens HPV-16, HPV-18, HPV-31 and HPV-45 were analyzed for cells expressing at least 2 of the following immune markers: CD40 Ligand, Interleukin-2, Tumor Necrosis Factor alpha or Interferon-gamma.
  An immune response is defined as 500 or more antigen-specific CD4 T-cells per million CD4 T-cells.
Time Frame: Day 0, Month 1 [Day 30], Month 7 and Month 18
Population: Analyses were performed on a subset (from pre-defined study sites) of subjects from the ATP cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 34 | 26
Participants
  HPV-16, Day 0: number analyzed (Participants) | 33 | 25
  HPV-16, Day 0 | 24 | 0
  HPV-16, Month 1: number analyzed (Participants) | 34 | 24
  HPV-16, Month 1 | 25 | 5
  HPV-16, Month 7: number analyzed (Participants) | 30 | 26
  HPV-16, Month 7 | 22 | 16
  HPV-16, Month 18: number analyzed (Participants) | 34 | 25
  HPV-16, Month 18 | 23 | 13
  HPV-18, Day 0: number analyzed (Participants) | 33 | 25
  HPV-18, Day 0 | 17 | 1
  HPV-18, Month 1: number analyzed (Participants) | 34 | 24
  HPV-18, Month 1 | 24 | 3
  HPV-18, Month 7: number analyzed (Participants) | 30 | 26
  HPV-18, Month 7 | 21 | 13
  HPV-18, Month 18: number analyzed (Participants) | 34 | 25
  HPV-18, Month 18 | 20 | 8
  HPV-31, Day 0: number analyzed (Participants) | 33 | 25
  HPV-31, Day 0 | 20 | 1
  HPV-31, Month 1: number analyzed (Participants) | 34 | 24
  HPV-31, Month 1 | 24 | 3
  HPV-31, Month 7: number analyzed (Participants) | 30 | 26
  HPV-31, Month 7 | 19 | 12
  HPV-31, Month 18: number analyzed (Participants) | 34 | 25
  HPV-31, Month 18 | 22 | 10
  HPV-45, Day 0: number analyzed (Participants) | 33 | 25
  HPV-45, Day 0 | 15 | 1
  HPV-45, Month 1: number analyzed (Participants) | 34 | 24
  HPV-45, Month 1 | 24 | 2
  HPV-45, Month 7: number analyzed (Participants) | 30 | 26
  HPV-45, Month 7 | 16 | 11
  HPV-45, Month 18: number analyzed (Participants) | 34 | 25
  HPV-45, Month 18 | 20 | 5

8. Secondary Outcome: Number of Subjects With Cluster of Differentiation 8 (CD8) T Cell-mediated Immune Responses Specific to Defined Oncogenic HPV Types
Description: CD8 T cell-mediated immune responses against the antigens HPV-16, HPV-18, HPV-31 and HPV-45 were analyzed for cells expressing at least 2 of the following immune markers: CD40 Ligand, Interleukin-2, Tumor Necrosis Factor alpha or Interferon-gamma.
  An immune response is defined as 200 or more antigen-specific CD8 T-cells per million CD8 T-cells.
Time Frame: Day 0, Month 1 [Day 30], Month 7 and Month 18
Population: Analyses were performed on a subset (from pre-defined study sites) of subjects from the ATP cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 34 | 25
Participants
  HPV-16, Day 0 | 0 | 0
  HPV-16, Month 1 | 1 | 0
  HPV-16, Month 7 | 0 | 2
  HPV-16, Month 18 | 1 | 0
  HPV-18, Day 0 | 0 | 0
  HPV-18, Month 1 | 0 | 1
  HPV-18, Month 7 | 0 | 1
  HPV-18, Month 18 | 1 | 0
  HPV-31, Day 0 | 0 | 0
  HPV-31, Month 1 | 0 | 0
  HPV-31, Month 7 | 2 | 1
  HPV-31, Month 18 | 1 | 0
  HPV-045, Day 0 | 0 | 0
  HPV-45, Month 1 | 0 | 1
  HPV-45, Month 7 | 2 | 0
  HPV-45, Month 18 | 0 | 0

9. Secondary Outcome: Number of Subjects With B Cell-mediated Immune Responses Specific to Defined Oncogenic HPV Types
Description: B-cell-mediated immune responses against the antigens HPV-16, HPV-18, HPV-31 and HPV-45 were measured by Enzyme-linked immunosorbent spot (ELISPOT) assay.
  A memory B-cell immune response was defined as presence of any antigen-specific memory B-cells per million B-cells.
Time Frame: Day 0, Month 1 [Day 30], Month 7 and Month 18
Population: Analyses were performed on a subset (from pre-defined study sites) of subjects from the ATP cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 34 | 26
Participants
  HPV-16, Day 0: number analyzed (Participants) | 33 | 25
  HPV-16, Day 0 | 20 | 1
  HPV-16, Month 1: number analyzed (Participants) | 34 | 24
  HPV-16, Month 1 | 27 | 21
  HPV-16, Month 7: number analyzed (Participants) | 30 | 26
  HPV-16, Month 7 | 26 | 20
  HPV-16, Month 18: number analyzed (Participants) | 34 | 25
  HPV-16, Month 18 | 17 | 11
  HPV-18, Day 0: number analyzed (Participants) | 33 | 25
  HPV-18, Day 0 | 21 | 3
  HPV-18, Month 1: number analyzed (Participants) | 34 | 24
  HPV-18, Month 1 | 27 | 18
  HPV-18, Month 7: number analyzed (Participants) | 30 | 26
  HPV-18, Month 7 | 26 | 20
  HPV-18, Month 18: number analyzed (Participants) | 34 | 25
  HPV-18, Month 18 | 18 | 15
  HPV-31, Day 0: number analyzed (Participants) | 33 | 25
  HPV-31, Day 0 | 20 | 1
  HPV-31, Month 1: number analyzed (Participants) | 34 | 24
  HPV-31, Month 1 | 24 | 3
  HPV-31, Month 7: number analyzed (Participants) | 30 | 26
  HPV-31, Month 7 | 21 | 15
  HPV-31, Month 18: number analyzed (Participants) | 34 | 25
  HPV-31, Month 18 | 11 | 6
  HPV-45, Day 0: number analyzed (Participants) | 33 | 25
  HPV-45, Day 0 | 15 | 1
  HPV-45, Month 1: number analyzed (Participants) | 34 | 24
  HPV-45, Month 1 | 24 | 2
  HPV-45, Month 7: number analyzed (Participants) | 30 | 26
  HPV-45, Month 7 | 18 | 11
  HPV-45, Month 18: number analyzed (Participants) | 34 | 25
  HPV-45, Month 18 | 14 | 6

10. Secondary Outcome: Number of Subjects Seropositive for Anti-HPV-16 and Anti-HPV-18 Antibodies in Cervico-vaginal Secretion Samples
Description: Seropositivity was defined as the detection of antibody titers above the limit of quantification by Enzyme-Linked Immunosorbant Assay. Defining a cut-off is technically not possible for this assay.
  Analyses were done in all collected samples from the evaluable subjects who provided cervical samples, with < 200 erythrocytes per microliter.
Time Frame: Day 0, Month 1 (Day 30), Month 7 and Month 18
Population: Analysis was performed on the subset of subjects from the ATP cohort for immunogenicity for whom cervical secretion samples were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 15 | 17
Participants
  Anti-HPV-16 Day 0: number analyzed (Participants) | 12 | 10
  Anti-HPV-16 Day 0 | 8 | 2
  Anti-HPV-16 Month 1: number analyzed (Participants) | 13 | 11
  Anti-HPV-16 Month 1 | 13 | 5
  Anti-HPV-16 Month 7: number analyzed (Participants) | 12 | 11
  Anti-HPV-16 Month 7 | 12 | 11
  Anti-HPV-16 Month 18 | 15 | 14
  Anti-HPV-18 Day 0: number analyzed (Participants) | 12 | 10
  Anti-HPV-18 Day 0 | 9 | 1
  Anti-HPV-18 Month 1: number analyzed (Participants) | 13 | 11
  Anti-HPV-18 Month 1 | 13 | 6
  Anti-HPV-18 Month 7: number analyzed (Participants) | 12 | 11
  Anti-HPV-18 Month 7 | 12 | 11
  Anti-HPV-18 Month 18 | 13 | 13

11. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies in Cervico-vaginal Secretion Samples
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
  Analyses were done in all collected samples from the evaluable subjects who provided cervical samples with < 200 erythrocytes per microliter.
Time Frame: Day 0, Month 1 (Day 30), Month 7 and Month 18
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 15 | 17
EL.U/mL
  Anti-HPV-16, Day 0: number analyzed (Participants) | 12 | 10
  Anti-HPV-16, Day 0 | 323.8 [84.0 to 1247.3] | 147.0 [93.3 to 231.6]
  Anti-HPV-16, Month 1: number analyzed (Participants) | 13 | 11
  Anti-HPV-16, Month 1 | 562.1 [312.8 to 1010.3] | 331.2 [100.3 to 1093.6]
  Anti-HPV-16, Month 7: number analyzed (Participants) | 12 | 11
  Anti-HPV-16, Month 7 | 220.5 [104.7 to 464.7] | 299.2 [153.4 to 583.3]
  Anti-HPV-16, Month 18 | 110.9 [46.2 to 266.0] | 52.8 [34.3 to 81.4]
  Anti-HPV-18, Day 0: number analyzed (Participants) | 12 | 10
  Anti-HPV-18, Day 0 | 177.1 [43.6 to 719.0] | 58.6 [58.6 to 58.6]
  Anti-HPV-18, Month 1: number analyzed (Participants) | 13 | 11
  Anti-HPV-18, Month 1 | 375.1 [257.8 to 545.8] | 54.0 [10.1 to 288.5]
  Anti-HPV-18, Month 7: number analyzed (Participants) | 12 | 11
  Anti-HPV-18, Month 7 | 111.5 [57.1 to 217.7] | 178.0 [88.0 to 359.9]
  Anti-HPV-18, Month 18 | 73.6 [31.2 to 173.4] | 29.6 [16.0 to 54.8]

12. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site.
  Solicited symptoms reported after the 4th vaccine dose in the 4-dose Group and across the 3 doses administered during this study in the 3-dose Group are disclosed.
Time Frame: Within 7 days after vaccination
Population: Analysis was performed on those subjects from the Total Vaccinated Cohort with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 64 | 48
Participants
  Pain | 61 | 45
  Redness | 24 | 18
  Swelling | 22 | 16

13. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, fever, gastrointestinal discomfort, headache, myalgia, rash and urticaria.
  Solicited symptoms reported after the 4th vaccine dose in the 4-dose Group and across the 3 doses administered during this study in the 3-dose Group are disclosed.
Time Frame: Within 7 days of vaccination
Population: Analysis was performed on those subjects from the Total Vaccinated Cohort with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 64 | 48
Participants
  Arthralgia | 10 | 4
  Fatigue | 33 | 33
  Fever (Oral or Axillary) ≥ 37.5 degrees Celsius | 4 | 5
  Gastrointestinal | 16 | 16
  Headache | 32 | 31
  Myalgia | 30 | 21
  Rash | 0 | 2
  Urticaria | 2 | 2

14. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An unsolicited adverse event is defined as any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
  AEs reported after the 4th vaccine dose in the 4-dose Group and after the 3 doses administered in this study in the 3-dose Group are disclosed.
Time Frame: Within 30 days of vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 65 | 50
Participants | 24 | 25

15. Secondary Outcome: Outcome of Any Reported Pregnancies
Description: Information on any subject who became pregnant while participating in this study was collected. The outcomes of the pregnancies are reported below.
Time Frame: From Day 0 up to Month 18
Population: Analysis was performed on those subjects reporting pregnancy during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 11 | 6
Participants
  Total number of pregnancies | 11 | 6
  Elective termination | 0 | 2
  Premature birth | 2 | 0
  Live infant | 8 | 4
  Pregnancy ongoing | 1 | 0

16. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs), New Onset of Autoimmune Diseases (NOADs) and Medically Significant Conditions (MSCs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies. MSC include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 up to Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 65 | 50
Participants
  NOCDs | 2 | 4
  NOADs | 0 | 2
  MSCs | 16 | 19

17. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Number analyzed (Participants) | 65 | 50
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited adverse events: from Day 0 to Day 6. Unsolicited adverse events: from Day 0 to Day 29. NOCDs, NOADs and MSCs: from Day 0 to Month 18.
Description: Events collected by systematic assessment are reported for subjects with a symptom diary card available.Events collected by non-systematic method are reported for the Total Vaccinated Cohort
Arm/Group | Cervarix™ 4-Dose Group | Cervarix™ 3-Dose Group
Serious Adverse Events (participants affected / at risk) | 1/65 | 1/50
Other Adverse Events (participants affected / at risk) | 62/65 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix™ 4-Dose Group (N=65) | Cervarix™ 3-Dose Group (N=50)
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix™ 4-Dose Group (N=65) | Cervarix™ 3-Dose Group (N=50)
Dizziness (Nervous system disorders) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Arthralgia (General disorders) | 10/64 | 4/48
Fatigue (General disorders) | 33/64 | 33/48
Fever (General disorders) | 4/64 | 5/48
Gastrointestinal symptoms (General disorders) | 16/64 | 16/48
Headache (General disorders) | 32 | 31/48
Myalgia (General disorders) | 30 | 21/48
Pain (General disorders) | 61/64 | 45/48
Redness (General disorders) | 24/64 | 18/48
Swelling (General disorders) | 22/64 | 16/48
Chlamydial infection (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.